CLINICAL TRIAL: NCT05731271
Title: A First-in-Human, Open-Label, Multi-Center Phase 1 Study of TST003 in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A First-in-Human, Phase 1 Study of TST003 in Subjects With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TST003-1001
Record Dates: First submitted 2023-01-05; First posted 2023-02-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Tumor; Colorectal Adenocarcinoma
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Interventional Model: Sequential Assignment Interventional Model Description: Bayesian Optimal Interval (BOIN) design followed by evaluation for efficacy and safety of TST003 as monotherapy at the recommended dose for dose expansion phase or RP2D in subjects with locally advanced or metastatic colorectal cancer (CRCMasking: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a Part - TST003 Dose Escalation (Experimental): TST003 administered every 3 weeks at increasing doses
  1 mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg, 30 mg/kg
  Interventions: Drug: TST003
- Phase 1b Part - Dose Expansion at Recommended Phase 2 dose (Experimental): Administer TST003 every 3 weeks to patients with positive GREM1 tumor expression at the recommended Phase 2 Dose,
  Interventions: Drug: TST003

INTERVENTIONS:
Drug: TST003 — IV humanized anti-GREM1 monoclonal antibody

SUMMARY:
The goal of this clinical trial is to test the safety of TST003 in patients with cancer.

The main question[s] it aims to answer are:

* What is the recommended dose patients can safely receive?
* How long does this drug remain in the body after administration?
* What are the side effects of this drug?
* Does your cancer respond to TST003?
* Participants on this study will get TST003 intravenously (through a needle into your vein), once every 3 weeks.
* You may need to come to the study site 2-4 times to have tests to see if you are eligible to be in the study before you begin to receive the study drug.
* After you start the study drug, you will need to return to the site several times after each dose so the physician can take vital signs, draw blood samples, and evaluate you for safety and wellbeing.
* Participants will continue taking the drug as long as they are receiving clinical benefit.
* At the end of your study participation, additional testing is required.

DETAILED DESCRIPTION:
Part 1 of the trial will consist cohorts, one dosed every 3 weeks at increasingly higher doses following the Bayesian Optimal Interval (BOIN) design. Part 1 is the dose finding portion of the trial. All locally advanced or metastatic solid tumors are accepted.

18 - 39 patients will be enrolled.

Part 2 consists of 2 pharmacodynamic cohorts of approximately 26-36 patients respectively. For Part 2, participants must have locally advanced or metastatic colorectal cancer (CRC).

The trial will last approximately 3 years, with assessments including but not limited to safety labs, ECGs, ECHO/MUGA, PKs and PDs and CT/MRI tumor assessments, and tumor biopsies based on emerging data found in Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of informed consent.
2. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.
3. Part 1: Subjects with histological or cytological diagnosed unresectable locally advanced or metastatic malignant solid tumors and who can provide archival tumor tissue. For Part 2: Subjects with histological or cytological diagnosed unresectable locally advanced or metastatic CRC and who can provide archival tumor tissue
4. Subjects who have tumor progression during or after prior therapy and for whom no standard therapy exists that would confer clinical benefit.
5. At least 1 measurable lesion per RECIST v1.1 ( Part 2 only).
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Life expectancy of 12 weeks or more.
8. Calculated creatinine clearance ≥30 mL/min per the Cockcroft and Gault formula. 9.Adequate bone marrow function:

   * Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 ×103/L);
   * Platelets ≥ 100,000/mm3 (≥ 100 × 109/L);
   * Hemoglobin ≥ 9.0 g/dL;

10.Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) ≤ 1.5 and Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 ULN (unless subjects are receiving therapeutic anti-coagulation which affects these parameters, and patients receiving therapeutic anticoagulation should be on a stable dose).

11.Adequate liver function as evidenced by bilirubin ≤1.5 × ULN and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN.

12.Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception during the treatment period and for at least 90 days after the last dose of TST003. Contraception methods should be consistent with local regulations.

Exclusion Criteria:

1. Untreated or symptomatic central nervous system (CNS) metastases. Note: Subjects with asymptomatic treated CNS metastases are eligible provided they have been clinically stable and not requiring steroid for at least 4 weeks following CNS -directed therapy are eligible for study entry.
2. Prior systemic anti-cancer treatment (chemotherapy, immunotherapy, biologic therapy, or targeted therapy or herbal medicine) within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose of study drug.
3. Radical radiation or local-regional therapies (transarterial chemoembolization or radiofrequency ablation) within 4 weeks prior to the first dose of study drug; palliative radiotherapy to a non-target lesion within 2 weeks prior to of study drug.
4. Any unresolved Grade 2 or greater toxicity from previous anticancer therapy except alopecia.
5. Any herbal medicine without anti-tumor intent within one week before the first dose of study drug.
6. History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases, including but not limited to pulmonary fibrosis, active pneumonitis.
7. Severe cardiovascular disease, including cerebrovascular accident, transient ischemic attack, myocardial infarction, or unstable angina, New York Heart Association (NYHA) class III or IV heart failure or uncontrolled arrhythmia within 6 months of the first dose.
8. Has the average corrected QT interval by Fridericia's formula (QTcF) prolongation to > 480 millisecond (ms) based on 12-lead ECG in triplicate, or with a history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives).
9. Uncontrolled hypertension (systolic pressure >150mmHg or diastolic pressure > 90mmHg).
10. Severe intestinal disease, including but not limited to:

    1. Peptic ulcer disease in the past 3 months prior to the first dosing.
    2. Clinically significant gastrointestinal bleeding as evidenced by hematemesis, hematochezia, or melena in the past 3 months prior to the first dosing without evidence of resolution documented by endoscopy or colonoscopy.
    3. Active colitis requiring ongoing treatment within 4 weeks prior to the first dosing, including infectious colitis, radiation colitis and ischemic colitis.
    4. History of ulcerative colitis or Crohn's disease.
11. Active or uncontrolled infections requiring IV of antibiotics, antivirals, or antifungals.
12. Active viral (any etiology) hepatitis except with the viral load below the limit quantification (hepatitis B virus (HBV) deoxyribonucleic acid (DNA) < 1000 copies/mL or 200 IU/mL; hepatitis C virus (HCV) ribonucleic acid (RNA) below the limit of quantification).
13. Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome.
14. Females who are pregnant or nursing.
15. Has known hypersensitivity to either the drug substances or inactive ingredients in the drug product.
16. Prior severe hypersensitivity to other antibodies, which in the opinion of the Investigator suggests an increased potential for hypersensitivity to study drug.
17. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks prior to the first dose of study drug.
18. Has a history or current evidence of any severe condition, concurrent therapy (e.g., psychiatric, substance abuse), or laboratory abnormality that might confound the interpretation of the study results, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the investigator.

    Additional Exclusion Criteria for Part 2 only (for Pharmacodynamic Cohorts)
19. Prior treatment with a GREM1 targeted therapy.
20. Any malignancy within 3 years prior to the first dosing of study drug except adequately treated localized carcinomas where standard therapy has been administered and patient is considered cured.
21. Subject will not be able to undergo on-treatment tumor biopsy on C3D1 per investigator's best judgement as baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assess the Dose limiting toxicities of TST003 | Observed during the first 21 day cycle
  Assess the Dose limiting toxicities experienced
Assess Adverse events (AEs) of TST003 | through study completion, an average of 1 year
  Assess Adverse events (AEs) as characterized by nature, frequency, and severity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Assess abnormal findings related to TST003 | through study completion, an average of 1 year
  Assess the abnormal findings of vital sign, physical examination, laboratory measurements, electrocardiogram (ECG) and echocardiogram (ECHO)/ multigated acquisition scan (MUGA) parameters
assess the Overall Response Rate of TST003 as monotherapy at the RP2D in subjects with locally advanced or metastatic GREM1 positive solid tumors (Phase 1bPart) | through study completion, an average of 1 year
  Overall Response Rate
assess the Duration of Response of TST003 as monotherapy at the RP2D in subjects with locally advanced or metastatic GREM1 positive solid tumors (Phase 1bPart) | through study completion, an average of 1 year
  Duration of Response
assess the Time to Response of TST003 as monotherapy at the RP2D in subjects with locally advanced or metastatic GREM1 positive solid tumors (Phase 1bPart) | through study completion, an average of 1 year
  Time to Response
assess the Disease Control Rate of TST003 as monotherapy at the RP2D in subjects with locally advanced or metastatic GREM1 positive solid tumors (Phase 1bPart) | through study completion, an average of 1 year
  Disease Control Rate
assess the Progression Free Survival of TST003 as monotherapy at the RP2D in subjects with locally advanced or metastatic GREM1 positive solid tumors (Phase 1bPart) | through study completion, an average of 1 year
  Progression Free Survival
assess the Overall Survival of TST003 as monotherapy at the RP2D in subjects with locally advanced or metastatic GREM1 positive solid tumors (Phase 1bPart) | through study completion, an average of 1 year
  Overall Survival Based on investigators' assessment using RECISTv1.1

SECONDARY OUTCOMES:
To characterize Area under the Curve (AUC) of TST003 | through study completion, an average of 1 year
  Determine AUC of serum concentration of TST003 over time
To characterize Cmax of TST003 | Measured while the patient is on study
  Determine Cmax of serum concentration of TST003
To Determine Trough serum concentration of TST003 | through study completion, an average of 1 year
  Determine Trough serum concentration of TST003
Determine the formation of Anti-drug antibody (ADA) against TST003 | through study completion, an average of 1 year
  Determine the formation of Anti-drug antibody (ADA) against TST003
Determine the formation of Neutralizing antibodies (NAb) against TST003 | through study completion, an average of 1 year
  Determine the formation of Neutralizing antibodies (NAb) against TST003

OTHER OUTCOMES:
To assess biomarkers in tumor tissue , and the correlation between biomarkers and PK, pharmacodynamic and clinical outcomes of TST003 | through study completion, an average of 1 year
  Analyze for biomarkers in tumor tissue samples including but not limited to GREM1, BMPs and FGFR1
To assess biomarkers, in blood and the correlation between biomarkers and PK, pharmacodynamic and clinical outcomes of TST003 | through study completion, an average of 1 year
  Analyze for biomarkers in blood samples including but not limited to GREM1 and BMPs

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - OHSU, Portland, Oregon
  - Mary Crowley, Dallas, Texas
  - NEXT Oncology, San Antonio, Texas